CLINICAL TRIAL: NCT06563843
Title: Comparison Between Velys Robotic-Assisted Solution (VRAS) and Conventional Surgery in Total Knee Arthroplasty: An Operational Excellence Evaluation
Brief Title: VRAS (Velys Robot-Assisted Solution) Operational Excellence Study
Status: Recruiting | Type: Observational
Sponsor: DEO NV (Industry)
Responsible Party: Sponsor
Other Study IDs: VRAS
Record Dates: First submitted 2024-07-17; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Total Knee Arthroplasty (TKA)
Keywords: VELYS; Total Knee Arthroplasty (TKA); Process flow; Robotic-assisted surgery; Operational excellence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Performing VELYS robot-assisted TKA: Surgeons performing VELYS robot-assisted TKA
  Interventions: Procedure: Robotic-assisted TKA
- Performing conventional TKA: Surgeons performing conventional TKA
  Interventions: Procedure: Conventional TKA

INTERVENTIONS:
Procedure: Robotic-assisted TKA — Robotic-assisted Total Knee Arthroplasty or total knee replacement is a surgical procedure using a robot to resurface a knee joint damaged with arthritis, and where the knee joint of the patient is replaced with a prosthesis.
  Other Names: DePuy Synthes, Velys Robotic-Assisted Solution
  Groups: Performing VELYS robot-assisted TKA
Procedure: Conventional TKA — Conventional Total Knee Arthroplasty or total knee replacement is a surgical procedure to manually resurface a knee joint damaged with arthritis, and where the knee joint of the patient is replaced with a prosthesis.
  Other Names: DePuy Synthes, Attune Knee System, Sigma Total Knee System
  Groups: Performing conventional TKA

SUMMARY:
The aim of this study is to investigate the differences in process set-up, efficiency, OR team workload, instrument trays and OR financial performance when using the VRAS (Velys Robotic Assisted Solution) of DePuy Synthes compared to conventional TKA.

DETAILED DESCRIPTION:
The increasing number of total knee arthroplasty (TKA) procedures is putting a significant burden on healthcare systems, surgeons and their surgical teams. Technology is introduced to improve accuracy, reproducibility and efficiency of TKA surgery, and a significant portion of the patient population is now being treated using Robotic Assisted Surgery. However, robotic surgeries are believed to have a longer procedure time.

The aim of this study is to investigate the differences in process set-up, efficiency, OR team workload, instrument trays and OR financial performance when using the VRAS (Velys Robotic Assisted Solution) of DePuy Synthes compared to conventional TKA.

In this multicentre study, measurements will be conducted in 10 hospitals with 10 selected surgeons across selected countries in Europe and the UK. For each surgeon enrolled, a minimum of five VRAS assisted surgical procedures and five conventional surgical procedures will be observed. The OR set-up will be similar for all cases in the same hospital. The same experienced surgeon will conduct all procedures.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic surgeons performing conventional and robot-assisted TKA

Exclusion Criteria:

* /

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The 10 participants of the study are orthopaedic surgeons. They will execute at least 5 conventional TKA procedures and at least 5 VELYS robot-assisted TKA procedures.
  This study is observational, with a focus on operational excellence, and as such DEO.care will not influence surgeon's decisions with regards to surgical technique philosophies. Surgeon will select the relevant techniques for each case at his/her own discretion.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-08-27 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Operational efficiency | 3 months
  Efficiency will be assessed using OR time, by comparing the OR days and procedures where TKR is performed conventionally or by using VRAS surgery.
  A granular analysis from the timestamps will be conducted using standard descriptive statistics. Additionally, the impaction process will be further analyzed, broken down into parts.

SECONDARY OUTCOMES:
Ergonomic impaction - weight of trays | 3 months
  Weight of trays will be measured to report ergonomic impaction of the team for the VRAS TKR compared to conventional TKR.
Ergonomic impaction - posture assessment | 3 months
  Surgeon's posture assessment using RULA and REBA method will be executed to report ergonomic impaction for the VRAS TKR compared to conventional TKR.
Total procedure cost | 3 months
  The procedure cost differences between VRAS TKR and conventional TKR will be calculated using activity based costing modeling. This model will include fixed direct, fixed indirect, and variable costs, tailored to each country's local cost parameters and healthcare financing models.

CONTACTS AND LOCATIONS:
Overall Officials: Willem Franssen, Msc., Study Director — DEOcare; Benjamin Bloch, M.D., Principal Investigator — Circle Health Group - BMI The Park Hospital
Locations (1):
- Circle health group - BMI The Park hospital, Nottingham, NG5 8RX, United Kingdom

IPD SHARING:
Plan to Share IPD: No